CLINICAL TRIAL: NCT06370039
Title: Phase 2, Multicenter, Randomized, Double-Masked, Vehicle-Controlled Study of INV-102 Ophthalmic Solution in Adult Subjects With Moderate to Severe Dry Eye Disease
Brief Title: Study of INV-102 Ophthalmic Solution in Adults With Moderate to Severe Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Invirsa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV-102-CS-003
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye; Keratoconjunctivitis sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INV-102 (Experimental): INV-102 0.7% ophthalmic solution administered for 4 weeks (twice daily [BID] for 2 weeks, then once daily [QD] for an additional 2 weeks)
  Interventions: Drug: INV-102
- Vehicle (Placebo Comparator): Vehicle ophthalmic solution administered for 4 weeks (BID for 2 weeks, then QD for an additional 2 weeks)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: INV-102 — INV-102 Ophthalmic Solution
  Arms: INV-102
Drug: Vehicle — Vehicle Ophthalmic Solution
  Arms: Vehicle

SUMMARY:
Phase 2 study to assess the efficacy of topically administered eyedrops of INV-102 during 4-week repeat dosing in subjects with moderate to severe dry eye disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects ≥18 and <75 years of age
* Presence of moderate to severe dry eye disease (DED) in at least one eye

Key Exclusion Criteria:

* Presently using prescription eyedrops, except those used for dry eye disease, which must be discontinued 4 weeks prior
* Use of over-the-counter (OTC) eyedrops except for lubricant eyedrops or artificial tears, within 1 week prior to initiation of study drug dosing
* History or evidence of ocular infection within the previous 30 days
* Blepharitis or meibomian gland disease requiring the use of either topical or systemic antibiotics within 2 months
* Allergic conjunctivitis requiring treatment within 30 days
* Unable to discontinue contact lens wear for 2 weeks prior and for the duration of the study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in corneal fluorescein staining total score on the National Eye Institute (NEI)/Industry scale | Baseline to Day 29
  Corneal fluorescein staining assessment will be performed using the NEI grading system to score each of 5 corneal zones (central, superior, lateral, medial, inferior) on a 0 to 3 scale (with a total score of 0 to 15). Higher scores indicate more corneal damage.

SECONDARY OUTCOMES:
Percentage of eyes with complete clearing of central corneal fluorescein staining | Baseline to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shalwitz, MD, Study Chair — Invirsa, Inc.
Locations (1):
- iuvo BioScience, Rush, New York, United States